CLINICAL TRIAL: NCT06976658
Title: Evaluating a Novel, Allosteric Glucokinase Activator in Monogenic Diabetes Secondary to Inactivating Glucokinase Mutations: a Randomised, Cross-over Trial
Brief Title: Glucokinase Activator in Monogenic Diabetes
Acronym: RESENSE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Elaine Chow, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RESENSE
Record Dates: First submitted 2025-03-22; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus; Monogenic Diabetes
Keywords: GCK-MODY; glucokinase activator
MeSH Terms: conditions — Diabetes Mellitus | interventions — Dorzagliatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigators, outcome assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): active drug or placebo in a cross over randomised sequence
  Interventions: Drug: Dorzagliatin
- placebo (Placebo Comparator): placebo in a cross over randomised sequence
  Interventions: Drug: matched placebo

INTERVENTIONS:
Drug: Dorzagliatin — Dorzagliatin 50mg bd
  Arms: Intervention
Drug: matched placebo — matched placebo
  Arms: placebo

SUMMARY:
Evaluating a novel, allosteric glucokinase activator in monogenic diabetes secondary to inactivating glucokinase mutations: a randomised, cross-over trial

DETAILED DESCRIPTION:
Evaluating a novel, allosteric glucokinase activator in monogenic diabetes secondary to inactivating glucokinase mutations: a randomised, cross-over trial

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and <75 years
2. body mass index (BMI) >18 and <30 kg/m2
3. fasting plasma glucose >5.6 mmol/L at screening
4. Participants with GCK-MODY had and are heterozygous carriers of a pathogenic or likely pathogenic GCK mutation at screening based on guidelines published by the American College of Medical Genetics and Genomics (ACMG), Association for Clinical Genomic Science (ACGS) and the ClinGen Monogenic Diabetes Expert Panel (MDEP) .

Exclusion Criteria:

1. Body weight <45kg at screening
2. Current or planning pregnancy or lactating
3. troke or cardiovascular disease within 6 months of recruitment
4. severe renal dysfunction (estimated glomerular filtration rate <30mL/min/1.73m2 or renal replacement therapy)
5. severe hepatic dysfunction (aspartate transaminase and/or alanine transaminase > 3 times upper limit of normal)
6. history of drug abuse or excessive alcohol intake
7. severe hypoglycemia within 6 months prior to screening
8. anaemia with Hb <10 g/dL at screening
9. excessive blood loss >300mL within 1 month of screening
10. use of strong or moderate CYP3A4 inhibitors or inducers
11. use of sulfonylureas, dipeptidyl peptidase-4 inhibitors, glucagon-like peptide-1 agonists, sodium glucose transporter 2 inhibitors, insulin, thiazolidinediones, acarbose in the 6 weeks prior to randomisation
12. use of long-term high-dose corticosteroids at randomisation
13. serious concurrent infections at time of screening

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose | 8 weeks
  Difference in fasting plasma glucose (FPG) between treatment periods

SECONDARY OUTCOMES:
• HbA1c | 8 weeks
  Difference between HbA1c at end of treatment periods
CGM metrics time in range | 8 weeks
  Time in range defined by CGM at end of treatment periods
CGM metric coefficient of variation | 8 weeks
  Difference in % CV at end of treatment periods
Glucose area under the curve during OGTT | 8 weeks
  Difference between AUC glucose at end of treament periods
Insulin area under the curve during OGTT | 8 weeks
  Difference between AUC insulin at end of treament periods
GLP1 area under the curve during OGTT | 8 weeks
  Difference between AUC GLP-1 at end of treament periods

OTHER OUTCOMES:
Treatment-emergent adverse events | 8 weeks
  Proportion of participants with adverse events in each treatment period
Hypoglycemia | 8 weeks
  Incidence of hypoglycemic events
Blood pressure | 8 weeks
  Blood pressure at end of each treatment period
Body weight | 8 weeks
  Body weight at end of each treatment period
Renal and liver function tests | 8 weeks
  Safety labs at end of treatment
Lipid profile | 8 weeks
  Safety labs at end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- 3M, Diabetes and Endocrine Research Center, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes